CLINICAL TRIAL: NCT04960020
Title: A New Etiological Cause for Anterior Cruciate Ligament Injury: E-Scooter
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Bulent KARSLIOGLU, Orthopedics and Traumatology specialist, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: E-scooter Related Injuries
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Anterior Cruciate Ligament Tear
Keywords: Anterior Cruciate Ligament injuries; e-scooter
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACL injuries with e-scooter trauma
  Interventions: Other: Retrospective Data Review

INTERVENTIONS:
Other: Retrospective Data Review — Retrospective Data Review

SUMMARY:
The investigators aimed to find the relationship between e-scooter use and anterior cruciate ligament injury.

DETAILED DESCRIPTION:
The incidence of injuries related to e-scooter use is increasing. There is no study in the literature investigating the relationship between anterior cruciate ligament injury and e-scooter use.

ELIGIBILITY:
Inclusion Criteria:

* Participants with e-scooter related ACL injury

Exclusion Criteria:

* Participants with other ACL injury etiology

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with e-scooter related ACL injury between January 2019-June 2021
Sampling Method: Probability Sample
Enrollment: 680 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Retrospective Evaluation | 2 years
  The investigators evaluated medical report of ACL injuried patients retrospectively

CONTACTS AND LOCATIONS:
Locations (1):
- SBU Prof. Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Li A, Zhao P, He H, Axhausen KW. Understanding the variations of micro-mobility behavior before and during COVID-19 pandemic period. Arbeitsberichte Verkehrs-und Raumplanung. 2020;1547.
- [Result] Kobayashi LM, Williams E, Brown CV, Emigh BJ, Bansal V, Badiee J, Checchi KD, Castillo EM, Doucet J. The e-merging e-pidemic of e-scooters. Trauma Surg Acute Care Open. 2019 Aug 29;4(1):e000337. doi: 10.1136/tsaco-2019-000337. eCollection 2019. PMID 31565677
- [Result] Tuncer S, Brown B. E-scooters on the ground: Lessons for redesigning urban micro-mobility. In: Proceedings of the 2020 CHI Conference on Human Factors in Computing Systems. 2020. p. 1-14.
- [Result] Trivedi TK, Liu C, Antonio ALM, Wheaton N, Kreger V, Yap A, Schriger D, Elmore JG. Injuries Associated With Standing Electric Scooter Use. JAMA Netw Open. 2019 Jan 4;2(1):e187381. doi: 10.1001/jamanetworkopen.2018.7381. PMID 30681711
- [Result] Stormann P, Klug A, Nau C, Verboket RD, Leiblein M, Muller D, Schweigkofler U, Hoffmann R, Marzi I, Lustenberger T. Characteristics and Injury Patterns in Electric-Scooter Related Accidents-A Prospective Two-Center Report from Germany. J Clin Med. 2020 May 22;9(5):1569. doi: 10.3390/jcm9051569. PMID 32455862
- [Result] Blomberg SNF, Rosenkrantz OCM, Lippert F, Collatz Christensen H. Injury from electric scooters in Copenhagen: a retrospective cohort study. BMJ Open. 2019 Dec 22;9(12):e033988. doi: 10.1136/bmjopen-2019-033988. PMID 31871261
- [Result] Ishmael CR, Hsiue PP, Zoller SD, Wang P, Hori KR, Gatto JD, Li R, Jeffcoat DM, Johnson EE, Bernthal NM. An Early Look at Operative Orthopaedic Injuries Associated with Electric Scooter Accidents: Bringing High-Energy Trauma to a Wider Audience. J Bone Joint Surg Am. 2020 Mar 4;102(5):e18. doi: 10.2106/JBJS.19.00390. PMID 31895168